CLINICAL TRIAL: NCT01329965
Title: Safety and Feasibility of an Endotoxemia Model: Pilot Study
Brief Title: Safety and Feasibility of an Endotoxemia Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PKE LPSpilot
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease; Inflammation
Keywords: Cardiovascular disease; Inflammation; LPS; Endotoxin
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LPS (Experimental): LPS will be injected at a dose of 0.6 ng/kg body weight through a catheter by a trained GCRC staff member involved with this study.
  Interventions: Drug: LPS (reference endotoxin, E. coli O113:H10:K:neg, manufactured under GMP)
- Saline (Placebo Comparator): A saline solution will be injected through a catheter by a trained GCRC staff member involved with this study.
  Interventions: Drug: LPS (reference endotoxin, E. coli O113:H10:K:neg, manufactured under GMP)

INTERVENTIONS:
Drug: LPS (reference endotoxin, E. coli O113:H10:K:neg, manufactured under GMP) — LPS or placebo (saline-salt water) will be injected (at approximately 7:30 am) in this catheter by a trained GCRC staff member involved with this study. Participants will not be told if they have received the drug or placebo. The LPS is a sterile solution of protein-free endotoxin which will be injected at a dose of 0.6 ng/kg body weight. Blood samples will be collected from a venous catheter for the first 12 hours and by venipuncture thereafter. Subjects will be continuously monitored by trained nursing staff for blood pressure (q 15 minutes) and body temperature (q 30 minutes), and the study will have physician oversight.

SUMMARY:
The purpose of this study is to establish the safety and feasibility of low dose LPS administration to a small subset of humans in preparation for a larger USDA funded study examining what is the lowest effective dose of EPA + DHA (300, 600, 900 and 1,800 mg/day delivered as fish oil supplements) that significantly attenuates the inflammatory response the investigators wish to examine the effects of an endotoxemia model for inducing inflammation. Based on previous research, low dose LPS administration affects metabolism in humans with only minimal clinical effects (such as "flu" like illness). Therefore, each of the six subjects included in this small pilot study will receive a low dose of LPS and placebo in order to learn more about the metabolic changes that occur during administration and inflammation. The investigators hypothesis that LPS administration will elicit only minimal clinical effects (such as "flu" like illness) when compared to placebo (saline--water with the same amount of salt as in your blood).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant/lactating women between the ages of 20 and 35 years old
* BMI > 19.9 and < 30.0
* Able to give written informed consent and willing to comply with all study- related procedures

Exclusion Criteria:

* Previous history of heart disease or diabetes
* Renal Insufficiency
* Chronic anti-inflammatory use
* Systolic blood pressure < 90
* Individuals currently using tobacco products or have done so in the previous 30 days
* Individuals taking Omega-3 fatty acid supplements or their usual intake of fish is greater than 3-4 servings per month

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory Markers | Baseline (before LPS administration), 1, 2, 3, 4, 6, 12, 24 hrs post LPS administration; 2, 3 and 5 days post LPS administration

SECONDARY OUTCOMES:
Change in Lipid Mediators | 1, 2, 3 and 5 days post LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States